CLINICAL TRIAL: NCT03683251
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of the Port Delivery System With Ranibizumab in Patients With Neovascular Age-Related Macular Degeneration (Portal)
Brief Title: Extension Study for the Port Delivery System With Ranibizumab (Portal)
Acronym: Portal
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR40549; 2020-004427-16 (EudraCT Number); 2023-507131-38-00 (EU CTIS Number)
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The sub-study 1 and sub-study 2 are open-label studies.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- PDS Implant Cohort 1 (US only) (Experimental): Participants with PDS implant from Study GX28228 treated with refill-exchanges of 100 mg/mL ranibizumab Q24W. Participants will switch to an every 12 weeks (Q12W) visit schedule from Week 168 to Week 240.
  Eligible participants from Study GX28228 will be enrolled upon completion of their final visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 2 (US only) (Experimental): Participants with PDS implant from Study GR40548 treated with refill-exchanges of 100 mg/mL ranibizumab Q24W. Participants will switch to an every 12 weeks (Q12W) visit schedule from Week 144 to Week 240.
  Eligible participants from Study GR40548 will be enrolled upon completion of their final visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 3 (US only) (Experimental): Participants in the intravitreal ranibizumab arm of Study GX28228 who will receive the PDS implant upon study entry and refill-exchanges of 100 mg/mL ranibizumab Q24W. Participants will switch to an every 12 weeks (Q12W) visit schedule from Week 168 to Week 240.
  Eligible participants from Study GX28228 will be enrolled upon completion of their final visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 4 (US only) (Experimental): Participants in the intravitreal ranibizumab arm of Study GR40548 who will receive the PDS implant upon study entry and refill-exchanges of 100 mg/mL ranibizumab Q24W. Participants will switch to an every 12 weeks (Q12W) visit schedule from Week 144 to Week 240.
  Eligible participants from Study GR40548 will be enrolled upon completion of their final visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 5 (ex-US only) (Experimental): Participants from Study WR42221 who completed Week 24 but were not eligible to be randomized within WR42221 and who will be treated with refill-exchanges of ranibizumab 100 mg/mL Q24W. Participants will be in the study for a minimum of 144 weeks and may continue after Week 144 until the PDS has received Health Authority approval (or non-approval) in their respective country and/or until the decision to close the study has been made by the sponsor.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 6 (ex-US only) (Experimental): Participants from Study WR42221 randomized to the Q24W arm, who will continue to be treated with refill-exchanges of ranibizumab 100 mg/mL Q24W. Participants will be in the study for a minimum of 144 weeks and may continue after Week 144 until the PDS has received Health Authority approval (or non-approval) in their respective country and/or until the decision to close the study has been made by the sponsor.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- PDS Implant Cohort 7 (ex-US only) (Experimental): Participants from Study WR42221 randomized to the Q36W arm, who will continue to be treated with refill-exchanges of ranibizumab 100 mg/mL Q36W. Participants will be in the study for a minimum of 144 weeks and may continue after Week 144 until the PDS has received Health Authority approval (or non-approval) in their respective country and/or until the decision to close the study has been made by the sponsor.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- Sub-study 1: PDS Implant (Experimental): Participants will receive PDS implant using TPC on Day 1 followed by refill-exchanges of ranibizumab 100 mg/mL via the PDS Q24W.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- Sub-study 2: Cohort 1 (Experimental): Participants will undergo re-implantation with the updated PDS implant and receive 2 refill-exchanges of ranibizumab 100 mg/mL Q24W.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- Sub-study 2: Cohort 2a (Experimental): Participants who received an updated PDS implant, have < 24 weeks post-re-implantation follow-up and no refill exchange visit in the main study, will undergo two refill-exchange procedures with ranibizumab 100 mg/mL Q24W post main study re-implantation visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL
- Sub-study 2: Cohort 2b (Experimental): Participants who received an updated PDS implant, have < 48 weeks post-re-implantation follow-up and one refill exchange visit in the main study, will undergo one refill-exchange procedure with ranibizumab 100 mg/mL Q24W post main study re-implantation visit.
  Interventions: Drug: PDS Implant with Ranibizumab 100 mg/mL

INTERVENTIONS:
Drug: PDS Implant with Ranibizumab 100 mg/mL — Will be administered as per the schedule described in individual arm

SUMMARY:
This study will evaluate the long-term safety and tolerability of the Port Delivery System with ranibizumab (PDS) (100 mg/mL) in participants with neovascular age-related macular degeneration (nAMD) who have either completed Phase II Study GX28228 (Ladder), Phase III Study GR40548 (Archway), Phase IIIb Study WR42221 (Velodrome), or completed Week 24 visit in Study WR42221 but were not eligible to be randomized in WR42221.

DETAILED DESCRIPTION:
The Transscleral Photocoagulation sub-study (sub-study 1) will evaluate the effectiveness of using transscleral photocoagulation (TPC) with the Iridex laser system to mitigate vitreous hemorrhages secondary to the Port Delivery System with ranibizumab (PDS) implantation procedure in participants with neovascular age-related macular degeneration (nAMD). The sub-study will enroll about 55 participants.

The Re-implantation sub-study (sub-study 2) will evaluate the safety of re-implantation with the updated PDS with ranibizumab . Up to 100 participants who previously participated in the main study in the United States will be enrolled and followed for a maximum of 72 weeks post-re-implantation in the substudy.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in and completion of Study GX28228 (Ladder) or Study GR40548 (Archway), without early treatment or study discontinuation in either study OR Previous enrollment in Study WR42221 (Velodrome) and either not eligible to be randomized in Study WR42221 at Week 24 or completed the study (from the Q24W or Q36W arm)
* Ability and willingness to undertake all scheduled visits and assessments
* For women of childbearing potential: agreement to remain abstinent or use contraceptive measures

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the treatment period and for at least 28 days after the last intravitreal injection of ranibizumab or 1 year after the last Implant refill-exchange of ranibizumab
* History of other ocular diseases that give reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab, that might affect interpretation of the results of the study or that renders the participant at high risk for treatment complications
* History of other diseases, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the Implant and that might affect interpretation of the results of the study or that renders the participant at high risk of treatment complications
* Requirement for continuous use of any medications or treatments indicated in the "Prohibited Therapy"

Sub-study 1

Inclusion Criteria

- For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures

Participants must meet the following ocular criteria for the study eye for substudy entry:

* Diagnosis of exudative nAMD within 2 years prior to the enrollment visit
* Previous treatment with at least two anti-VEGF ITV injections (e.g., ranibizumab, bevacizumab, or aflibercept) for nAMD per standard of care within 6 months prior to the enrollment visit
* Demonstrated response to prior anti-VEGF ITV treatment since diagnosis, as evidenced at enrollment by the following:

Overall decrease in nAMD disease activity detected on SD-OCT AND Stable or improved best-corrected visual acuity (BCVA)

* All subtypes of nAMD lesions are permissible (i.e., type I, type II, type III, or mixed forms per optical coherence tomography (OCT) classification) nAMD lesions at the time of diagnosis must involve the macula (6 mm diameter centered at the fovea).
* Sufficiently clear ocular media and adequate pupillary dilation to allow for analysis and grading by the central reading center of FP and SD-OCT images.

Exclusion Criteria Prior Ocular Treatments Study Eye

* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* Prior treatment with Visudyne, external-beam radiation therapy, or transpupillary thermotherapy
* Previous treatment with corticosteroid ITV injection
* Previous intraocular device implantation
* Previous laser (any type) used for AMD treatment

Either Eye

* Treatment with anti-VEGF agents other than ranibizumab within 1 month prior to the enrollment visit
* Prior participation in a clinical trial involving anti-VEGF drugs within 6 months prior to the enrollment visit, other than ranibizumab

CNV Lesion Charateristics Study Eye

* Subretinal hemorrhage that involves the center of the fovea, if the hemorrhage is greater than 0.5 disc area (1.27 mm2 ) in size at screening
* Subfoveal fibrosis or subfoveal atrophy

Either Eye

- CNV due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia

Concurrent Ocular Conditions Study Eye

* Retinal pigment epithelial tear
* Any concurrent intraocular condition (e.g., cataract, glaucoma, diabetic retinopathy, or epiretinal membrane) that would either require surgical intervention during the study to prevent or treat visual loss that might result from that condition or affect interpretation of study results
* Active intraocular inflammation (grade trace or above)
* History of vitreous hemorrhage
* History of rhegmatogenous retinal detachment
* History of rhegmatogenous retinal tears or peripheral retinal breaks within 3 months prior to the enrollment visit
* Aphakia or absence of the posterior capsule
* Previous violation of the posterior capsule is also an exclusion criterion unless it occurred as a result of yttrium-aluminum garnet (YAG) laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation.
* Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia
* Preoperative refractive error that exceeds 8 diopters of myopia, for participants who have undergone prior refractive or cataract surgery in the study eye
* Intraocular surgery (including cataract surgery) within 3 months preceding the enrollment visit
* Uncontrolled ocular hypertension or glaucoma and any such condition the investigator determines may require a glaucoma-filtering surgery during a patient's participation in the study
* History of glaucoma-filtering surgery, tube shunts, or microinvasive glaucoma surgery
* History of corneal transplant
* History of prior vitrectomy surgery and absence of posterior capsule

Either Eye

* History of idiopathic or autoimmune-associated uveitis
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis

Concurrent Systemic Conditions

* Inability to comply with study schedule or procedures as described in the study protocol
* Uncontrolled blood pressure
* History of stroke within the last 3 months prior to informed consent
* Uncontrolled atrial fibrillation within 3 months of informed consent
* History of myocardial infarction within the last 3 months prior to informed consent
* History of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of ranibizumab or placement of the implant and that might affect interpretation of the results of the study or renders the patient at high risk of treatment complications in the opinion of the investigator
* Current systemic treatment for a confirmed active systemic infection
* Use of any systemic anti-VEGF agents
* Chronic use of oral corticosteroids
* Active cancer within 12 months of enrollment
* Previous participation in any non-ocular (systemic) disease studies of investigational drugs within 1 month preceding the informed consent (excluding vitamins and minerals)
* Use of antimitotic or antimetabolite therapy within 30 days or 5 elimination half-lives of the enrollment visit
* History of albinism
* Pregnant or breastfeeding, or intending to become pregnant during the treatment period and for at least 28 days after the last ITV injection of ranibizumab or 1 year after the last implant refill-exchange of ranibizumab

Sub-study 2

Inclusion Criteria:

* Having experienced septum dislodgement in the original implant while in the main study or after exiting the main study Ocular Inclusion Criteria for Study Eye
* Sufficiently clear ocular media and adequate pupillary dilation to allow for analysis and grading by central reading center

Exclusion Criteria (Cohort 1 only):

Concurrent Ocular Conditions-Study Eye

* Any ocular condition that may render the patient at high risk for surgical or treatment complications
* Intraocular surgery (including cataract surgery) within 1 month preceding the enrollment visit
* Any use of medicated intraocular implants (other than the PDS implant), at any time prior to enrollment
* History of rhegmatogenous retinal tears or peripheral retinal breaks within 3 months prior to the enrollment visit
* Any concurrent ocular condition that would require surgical intervention during the study to prevent or treat visual loss
* Concurrent conjunctival, Tenon's capsule, and/or scleral condition in the supero-temporal quadrant of the eye (e.g., scarring, thinning, mass) that may affect the refill-exchange procedure of the PDS implant
* Ongoing ocular complications that might affect participant safety

Concurrent Ocular Conditions-Either Eye

* Suspected or active ocular or periocular infection
* Any history of uveitis
* Active blepharitis

Concurrent Systemic Conditions

* Recent history (in the last 3 months prior to enrollment) of other disease, other non-diabetic metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a condition that contraindicates the use of ranibizumab or surgical placement of the PDS implant; that might affect interpretation of the results of the study; or that renders the participant at high risk for treatment complications
* Active cancer within the last 12 months, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or prostate cancer
* Current systemic treatment for a confirmed active systemic infection - Participation in an investigational trial that involves treatment with any drug or device (with the exception of vitamins and minerals or enrollment in the main study GR40549) within 6 months prior to enrollment.
* Use of antimitotic or antimetabolite therapy within 30 days or 5 elimination half-lives.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Ocular and Systemic (Non-Ocular) Adverse Events (AEs) | Baseline up to Week 240
Incidence, Severity, and Duration of Adverse Event of Special Interest (AESIs) | Baseline up to Week 240
Incidence, Severity, and Duration of PDS-Associated Ocular AESIs During the Postoperative Period (Up to 37 days of Initial Implantation) and Follow-Up Period (>37 days After Implantation Surgery) for Participants who Receive the PDS Implant in the Study | Baseline up to Week 240
Incidence and Severity of Adverse Device Effects | Baseline up to Week 240
Incidence, Causality, Severity, And Duration Of Anticipated Serious Adverse Device Effects | Baseline up to Week 240
Sub-study 1: Rate of Vitreous Hemorrhage Secondary to Choroidal Bleeding That Does not Resolve by the Week 4 Visit After Implant Insertion Surgery. | Baseline to Week 4
Sub-study 2: Number of Participants with Ocular and Systemic (Non-ocular) Adverse Events (AEs) and Severity of These AEs | Baseline to Week 72
Sub-study 2: Number of Participants with Adverse Events of Special Interests (AESIs) and Severity of AESIs | Baseline to Week 72
Sub-study 2: Duration of AESIs | Baseline to Week 72
Sub-study 2: Number of participants with Ocular AESIs and Severity of Ocular AESIs During the Post-operative Period | Up to Day 37 post re-implantation
Sub-study 2: Number of participants with Ocular AESIs and Severity of Ocular AESIs During the Follow-up Period | > 37 days post re-implantation (up to approximately Week 72)
Sub-study 2: Duration of Ocular AESIs During the Post-operative Period | Up to Day 37 post re-implantation
Sub-study 2: Duration of Ocular AESIs During the Follow-up Period | > 37 days post re-implantation (up to approximately Week 72)
Sub-study 2: Number of Participants with Adverse Device Effects (ADEs) and Severity of ADEs | Baseline to Week 72
Sub-study 2: Number of Participants with Anticipated Serious ADEs and Severity of Anticipated Serious ADEs | Baseline to Week 72
Sub-study 2: Duration of Anticipated Serious ADEs | Baseline to Week 72
Sub-study 2: Number of Device Deficiencies | Baseline to Week 72

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) Score from Baseline Over Time, as Assessed using the ETDRS Visual Acuity Chart at a Starting Distance of 4 Meters | Baseline up to Week 240
  ETDRS = Early Treatment Diabetic Retinopathy Study
  A vision score of 20/20 vision is considered normal. A score of 20/200 is considered being legally blind.
Percentage of Participants who Lose <15, <10, or <5 Letters in BCVA Score from Baseline Over Time | Baseline up to Week 240
Percentage of Participants with BCVA Score of 38 Letters (of 20/200 Approximate Snellen Equivalent) or Worse over Time | Baseline up to Week 240
Percentage of Participants with BCVA Score of 69 Letters (20/40 Approximate Snellen Equivalent) or Better over Time | Baseline up to Week 240
Change from Baseline in Center Point Thickness (CPT) Over Time | Baseline up to Week 240
  CPT is defined as the retinal thickness in the center point of the fovea measured between the internal limiting membrane and the inner third of the retinal pigment epithelium layer. CPT is measured using optical coherence tomography (OCT).
Percentage of Participants who Undergo Supplemental Treatment with Intravitreal Ranibizumab 0.5 mg During Each Refill-exchange Interval | Baseline up to Week 240
Sub-study 1: Incidence of Ocular Adverse Events (AEs) and Adverse Events of Special Interest (AESIs) in the Study eye | Baseline up to Week 104
Sub-study 1: Incidence of AEs Commonly Seen After Transscleral Cyclophotocoagulation (TS-CPC) for Treatment of Glaucoma in the Study eye | Baseline up to Week 104
Sub-study 1: Time From Surgery to Vitreous Hemorrhage Resolution in the Study eye | Baseline up to Week 104
Sub-study 1: Incidence of Vitreous Hemorrhage Grade 3 and Higher in the Study eye over time | Baseline up to Week 104
Sub-study 1: Distribution of Vitreous Hemorrhage Grade in the Study eye Over Time | Baseline up to Week 104
Sub-study 1: Rate of Vitrectomy in the Study eye | Baseline up to Week 104
Sub-study 1: Percentage of Participants who Lose <15, <10, or <5 Letters in BCVA Score From Baseline Over Time | Baseline up to Week 104
Sub-study 1: Change in BCVA Score From Baseline Over Time | Baseline up to Week 104
Sub-study 1: Change from Baseline in CPT Over Time | Baseline up to Week 104
Sub-study 1: Change From Baseline in Center Subfield Thickness (CST) Over Time | Baseline up to Week 104
Sub-study 2: Number of Participants with Ocular AESIs and Severity of AESIs Following Refill-exchange | Up to approximately Week 72
Sub-study 2: Duration of AESIs Following Refill-exchange | Up to approximately Week 72
Sub-study 2: Number of Participants With ADEs and Severity of ADEs Following Refill-exchange | Up to approximately Week 72
Sub-study 2: Number of Participants with Anticipated Serious ADEs and Severity of Anticipated Serious ADEs Following Refill-exchange | Up to approximately Week 72
Sub-study 2: Number of Device Deficiencies Following Refill-exchange | Up to approximately Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (165):
- United States (81):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Jacobs Retina center at the Shiley eye Institute UCSD, La Jolla, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - N CA Retina Vitreous Assoc, Mountain View, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - UCSF, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - Southwest Retina Consultants, Durango, Colorado
  - Eye Center of Northern CO, Fort Collins, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Florida Eye Microsurgical Inst, Boynton Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Illinois Retina Associates, Joliet, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Retina Specialists, Towson, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC., Minneapolis, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - The Retina Institute - Chesterfield, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Retina Assoc of Western NY, Rochester, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Retina Vit Surgeons/Central NY, Syracuse, New York
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - OSU Eye Physicians & Surgeons, Columbus, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Retina Northwest, Portland, Oregon
  - Oregon HSU, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, Florence, South Carolina
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Med Center Ophthalmology Assoc, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Wagner Kapoor Institute, Virginia Beach, Virginia
  - Pacific Northwest Retina, Silverdale, Washington
  - Spokane Eye Clinical Research, Spokane, Washington
- Argentina (3):
  - Oftalmos, Capital Federal
  - Centro Oftalmologico Dr. Charles S.A., Ciudad Autonoma Buenos Aires
  - Grupo Laser Vision, Rosario
- Australia (2):
  - Eyeclinic Albury Wodonga, Albury, New South Wales
  - Eye and Retina Consultants, Hurstville, New South Wales
- Austria (2):
  - LKH-Univ.Klinikum Graz, Graz
  - Medizinische Universitat Wien, Vienna
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (5):
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Retina Clinic, São Paulo, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESPX, São Paulo, São Paulo
  - Instituto da Visao IPEPO, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- France (5):
  - Centre Retine Gallien, Bordeaux
  - Hopital de la croix rousse, Lyon
  - Centre Paradis Monticelli, Marseille
  - Hopital Lariboisiere, Paris
  - Fondation Rothschild, Paris
- Germany (12):
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinikum Koln, Cologne
  - Medizinische Universitat Lausitz ? Carl Thiem, Cottbus
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - LMU Klinikum der Universitat, Augenklinik, München
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitatsklinikum Munster, Münster
  - Knappschaftsklinikum Saar GmbH, Sulzbach
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Augenklinik und Poliklinik, Ulm
- Israel (6):
  - Rambam Medical Center, Haifa
  - Hadassah MC, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky MC, Tel Aviv
- Italy (13):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Policlinico di Bari, Bari, Apulia
  - Azienda Ospedaliero Universitaria "Ospedali Riuniti" Trieste-Ospedale Maggiore, Trieste, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena, Milan, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Asst Fatebenefratelli Sacco, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette - Ancona, The Marches
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia, Perugia, Umbria
  - Ospedale Classificato Equiparato Sacro Cuore ? Don Calabria, Negrar - Verona, Veneto
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Veneto
- Spain (12):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega, Oviedo, Principality of Asturias
  - Oftalvist Valencia, Burjassot, Valencia
  - Centro de Oftalmologia Barraquer, Barcelona
  - Institut de la Macula i la retina, Barcelona
  - Hospital dos de maig, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Arruzafa. Servicio de Oftalmologia, Córdoba
  - Clinica Baviera, Madrid
- Switzerland (5):
  - Universitatsspital Basel Augenklinik Klinik, Basel
  - Inselspital Bern Ophthalmologische Klinik, Bern
  - Vista Klinik Ophthalmologische Klinik, Binningen
  - Fondation Asile Des Aveugles ? Jules Gonin Eye Hospital, Lausanne
  - Stadtspital Triemli Ophthalmologische Klinik, Zurich
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
  - National Taiwan University Hospital, Zhongzheng Dist.
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Etlik City Hospital, Ankara
  - Beyoglu Goz Training and Research Hospital, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
- United Kingdom (8):
  - Bristol Eye Hospital, Bristol
  - Royal Liverpool University Hospital, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Central Middlesex Hospital, London
  - Kings College Hospital NHS Foundation Trust, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Sunderland Eye Infirmary, Sunderland
  - Royal Wolverhampton hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Eichenbaum DA, Freeman WR, Chang MA, Brooks L, Chaudhry N, Dadgostar H, McCannel CA, Michels M, Mittra RA, Wolfe JD, Beindl VC, Jaycock P, Bobbala A, Gune S, Spicer G, Callaway N. Endophthalmitis in Eyes Treated with the Port Delivery System with Ranibizumab: Summary of Cases during Clinical Trial Development. Ophthalmol Retina. 2025 Feb;9(2):127-143. doi: 10.1016/j.oret.2024.08.005. Epub 2024 Aug 16. PMID 39154860